CLINICAL TRIAL: NCT06271135
Title: Assessing the Quality of Life of Patients With Rosacea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Bialystok (Other)
Collaborators: University of Lomza (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LU20170508
Record Dates: First submitted 2024-02-06; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Rosacea
Keywords: quality of life; cosmetics procedures; lifestyle; dietary antioxidants
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with rosacea (Experimental)
  Interventions: Behavioral: CAPILLARY REPAIR SERUM 30ml

INTERVENTIONS:
Behavioral: CAPILLARY REPAIR SERUM 30ml — Cosmetic procedures were performed on a group of patients after a cosmetic interview containing questions about contraindications to the procedure. The treatment was performed 3-times at 2-week intervals and consisted of cavitation peeling and sonophore-sis with an antioxidant preparation dedicated to vascular skin. The F-808 Skin Scrubber device was used for the treatment. After a month, the procedure was repeated. The stages of a cosmetologist's procedure during a cosmetic intervention were as follows: 1. make-up removal; 2. skin diagnostics, exclusion of contraindications, discussion of the procedure; 3. cavitation peeling - gentle skin cleansing using ultrasound; 4. applying an antioxidant cosmetic mixture (composition: rutin, horse chestnut and arnica extract, acerola, vitamin C, moisturizing complex of algae); 5. performing sonophoresis treatment; 6. applying the cream at the end; 7. discussion of indications for further care.

SUMMARY:
The study population consisted of 160 patients (123 women and 37 men) with rosacea, who agreed to participate in this study. Patients were qualified for the study among people visiting the cosmetic studio in Choroszcz in the period from June 2017 to November 2018, based on the diagnosis of a dermatologist and cosmetologist. The cosmetic intervention was performed using CAPILLARY REPAIR SERUM (30ml). Study participants completed self-reported questionnaire and standardized questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* the inclusion criteria were: age ≥ 30 years,
* diagnosis of rosacea according to the criteria of the National Rosacea Society Expert Committee (NRSEC) from 2019,
* tolerance to the ingredients of the preparation used in the cosmetic intervention,
* lack of pregnancy and lactation,
* completion of a survey,
* signed informed consent

Exclusion Criteria:

* age < 30 years,
* patients with other facial skin diseases (e.g. acne, psoriasis, eczema),
* intolerance to the ingredients of the preparation used in the cosmetic treatment,
* patients with neuropsychiatric diseases, pregnancy, lactation,
* patients who did not sign informed consent to participate in the study
* did not complete the survey questionnaire.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Elements influenced on quality of life of participants with rosacea | 17 months
  The aim of the study was to assess whether antioxidant cosmetic procedures and selected lifestyle elements, especially dietary antioxidants have a significant impact on the quality of life of patients with rosacea.

SECONDARY OUTCOMES:
Self-reported questionnaire | 17 months
  Author's questionnaire containing questions on sociodemographic status, anthropometic data, health behaviors, lifestyle, and information on rosacea.
Dietary Questionnaire | 17 months
  Energy of diet and nutrients intake were assessed using 3-day 24-h dietary recalls (two randomly selected weekdays and one weekend day) and computer program Diet 6.0.
The Physical Activity Questionnaire | 17 months
  The physical activity was assessed by a short version of the International Physical Activity Questionnaire (IPAQ).
DLQI (Dermatology Life Quality Index) | 17 months
  The assessment of quality of life in rosacea was carried out using the Polish version of standardized questionnaire DLQI (Dermatology Life Quality Index).
SWLS (Satisfaction With Life Scale) | 17 months
  The assessment of satisfaction with life in patients with rosacea was carried out using the Polish version of standardized questionnaire SWLS (Satisfaction With Life Scale).
BDI (Beck Depression Inventory) | 17 months
  The assessment of depression in patients with rosacea was carried out using the Polish version of standardized questionnaire BDI (Beck Depression Inventory).

CONTACTS AND LOCATIONS:
Overall Officials: Małgorzata E Zujko, Dr., Principal Investigator — Medical Univeristy of Bialystok
Locations (1):
- Medical University of Bialystok, Bialystok, Poland